CLINICAL TRIAL: NCT04924335
Title: Ultrasound-guided Erector Spinae Plane (ESP) Block Attenuates Surgery-related Stress Response in Cardiac Surgery Patients Undergoing Enhanced Recovery After Surgery (ERAS) Program
Brief Title: The Effects of Erector Spinae Plane (ESP) Block on Surgery-related Stress Response in Cardiac Surgery With ERAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Eda Balci, Medical Doctor, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MH2.2
Record Dates: First submitted 2021-05-22; First posted 2021-06-14 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Surgery Stress
Keywords: erector spinae plane block; cardiac surgery; enhanced recovery after surgery program; lactate; stress response; c reactive protein
MeSH Terms: conditions — Fractures, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESP group (Active Comparator): ESP group patients will be performed ultrasound-guided erector spinae plane block with 20 ml 0.025% Bupivacaine, preoperatively and will receive ERAS cardiac anesthesia protocol
  Interventions: Procedure: Erector spinae plane block
- Conventional group (No Intervention): The conventional group will receive ERAS cardiac anesthesia protocol

INTERVENTIONS:
Procedure: Erector spinae plane block — Preoperative ultrasound-guided bilateral erector spinae plane block with 20 ml 0.025% bupivacaine.
  Arms: ESP group

SUMMARY:
Surgery-induced pain reveals its own metabolic and inflammatory responses, resulting in a further increase in noxious pathways that are already occurring. Even though it is difficult to distinguish whether the metabolic and inflammatory responses are pain-induced or surgical-induced, it is clear that pain can cause a response. This study aims to investigate the effects of erector spinae plane block on surgery-related stress response with enhanced recovery after cardiac surgery protocol.

DETAILED DESCRIPTION:
The Enhanced Recovery After Cardiac Surgery (ERAS Cardiac) program includes a perioperative multimodal, opioid-sparing pain management plan as an essential component of any comprehensive program. A multimodal pain management plan is nonopioid systemic analgesic agents, regional and local anesthetic techniques, and judicious use of opioids. This study aims to examine inflammatory and hematological parameters in patients who underwent cardiac surgery with ERAS, with and without preoperative bilateral erector spinae plane block (ESP). For this purpose, the presence of an obstacle ESP block application in the preoperative period will be investigated in patients who are prepared for cardiac surgery according to ERAS principles, and the patient's group will be determined accordingly. An analgesia protocol that does not include a regional technique will be applied to the patient in cases such as the patient's refusal to allow preoperative block and the presence of a situation that does not allow blockage in the block area. The perioperative characteristics of ERAS patients with and without ESP block will be examined, intraoperative lactate, and preop-postoperative hemogram-albumin-C reactive protein parameters will be recorded.

ERAS patients with ESP block: After preparation in accordance with the ERAS protocol, ultrasound-guided bilateral ESP block will be performed with 20 ml of 0.025% bupivacaine at T5-7 levels in patients taken to the operating room in the preoperative period, and will be administered intraoperative low-dose remifentanil infusion and sevoflurane anesthesia.

ERAS patients without ESP block: After preparation according to the ERAS protocol, patients will be administered lidocaine, ketamine, paracetamol, and intraoperative low-dose remifentanil infusion and sevoflurane anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who will undergo open-heart surgery with ERAS protocol

Exclusion Criteria:

* Emergency surgeries
* Patients with allergic reactions to anesthesia and analgesia drugs to be used
* Patients who do not want to participate in the study voluntarily
* Severe systemic disease (kidney, liver, pulmonary, endocrine)
* Substance abuse history
* History of chronic pain
* Psychiatric problems and communication difficulties
* Patients who need revision due to hemostasis in the postoperative period
* Patients with severe hemodynamic instability due to infection, heavy bleeding, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Basal measurements- after anesthesia induction | After anesthesia induction, an average of 5 minutes
  After induction of anesthesia, blood gas analysis will be performed and lactate level (mmol/L) will be recorded.
Basal measurements- after anesthesia induction | After anesthesia induction, an average of 5 minutes
  After induction of anesthesia, blood gas analysis will be performed and hemoglobin level (g/dL) will be recorded.
Second measurements- after cardiopulmonary bypass initiation | After cardiopulmonary bypass inititation, an average of 5 minutes
  After cardiopulmonary bypass initiation, blood gas analysis will be performed and lactate level (mmol/L) will be recorded.
Second measurements- after cardiopulmonary bypass initiation | After cardiopulmonary bypass inititation, an average of 5 minutes
  After cardiopulmonary bypass initiation, blood gas analysis will be performed and hemoglobin level (g/dL) will be recorded.
Third measurements- during cardiopulmonary bypass, at lowest temperature | During cardiopulmonary bypass, an average of 10 minutes
  During cardiopulmonary bypass, at lowest temperature, blood gas analysis will be performed and lactate level (mmol/L) will be recorded.
Third measurements- during cardiopulmonary bypass, at lowest temperature | During cardiopulmonary bypass, an average of 10 minutes
  During cardiopulmonary bypass, at lowest temperature, blood gas analysis will be performed and hemoglobin level (g/dL) will be recorded.
Fourth measurements- end of cardiopulmonary bypass | At the end of cardiopulmonary bypass, an average of 10 minutes
  At the end of cardiopulmonary bypass, blood gas analysis will be performed and lactate level (mmol/L) will be recorded.
Fourth measurements- end of cardiopulmonary bypass | At the end of cardiopulmonary bypass, an average of 10 minutes
  At the end of cardiopulmonary bypass, blood gas analysis will be performed and hemoglobin level (g(dL) will be recorded.
Fifth measurements- end of surgery | At the end of surgery, an average of 20 minutes
  At the end of surgery, blood gas analysis will be performed and lactate level (mmol/L) will be recorded.
Fifth measurements- end of surgery | At the end of surgery, an average of 20 minutes
  At the end of surgery, blood gas analysis will be performed and hemoglobin level (g/dL) will be recorded.

SECONDARY OUTCOMES:
Preoperative complete blood count | The day before surgery, 24 hours
  Preoperative complete blood count will be evaluated and recorded.
Preoperative albumin | The day before surgery, 24 hours
  Preoperative albumin levels will be evaluated and recorded.
Postoperative C reactive protein | 6 hours after surgery
  Postoperative C reactive protein levels will be evaluated and recorded.
Postoperative complete blood count | 6 hours after surgery
  Postoperative complete blood count will be evaluated and recorded.
Postoperative albumin | 6 hours after surgery
  Postoperative albumin levels will be evaluated and recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Serdar Günaydın, Professor, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara City Hospital, Ankara, Select State/Province, Turkey (Türkiye)